CLINICAL TRIAL: NCT06684171
Title: A Randomized Clinical Trial of Transcatheter Edge-to-edge Repair for Mitral Regurgitation Under Fully Echocardiographic Guidance Compared with Under Combined Guidance of Both Echocardiography and Fluoroscopy (ECHO-CLIP Study)
Brief Title: Comparison of Transcatheter Edge-to-edge Repair Using Echo Only with Echo Combined with X Ray for Mitral Regurgitation (ECHO-CLIP)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pan Xiangbin (Other)
Responsible Party: Sponsor-Investigator, Pan Xiangbin, The Vice President of Fuwai Hospital, Chinese Academy of Medical Sciences, and Director of the Structural Heart Disease Center., Chinese Academy of Medical Sciences, Fuwai Hospital
Organization: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NO.SP2024005(01)A
Record Dates: First submitted 2024-11-04; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Mitral Regurgitation
Keywords: mitral regurgitation; transcatheter edge-to-edge repair; ECHO-CLIP; randomized clinical trail; ultrasound; echo
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Echocardiography-guided group (Experimental): Patients randomized to the echocardiography-guided group will undergo TEER procedure under fully echo guidance.
  Interventions: Procedure: Echocardiographic guidance
- Fluoroscopy-guided group (Active Comparator): Patients randomized to the fluoroscopy-guided group will undergo TEER procedure under combined guidance of X ray and echo.
  Interventions: Procedure: Fluoroscopic guidance

INTERVENTIONS:
Procedure: Echocardiographic guidance — After detailed evaluation, patients randomized in this group will undergo TEER procedure under guidance of fully echocardiography but any fluoroscopy in the entire process.
  Arms: Echocardiography-guided group
Procedure: Fluoroscopic guidance — After detailed evaluation, patients randomized in this group will undergo TEER procedure under combined guidance of echocardiography and fluoroscopy in the entire process.
  Arms: Fluoroscopy-guided group

SUMMARY:
Mitral regurgitation (MR) is a common valvular heart disease in the elderly population, frequently associated with poor prognosis if not treated. Transcatheter edge-to-edge repair (TEER) has recently emerged as a popular strategy due to minimal invasiveness. What's more, previous studies, such as EVEREST II and COAPT study, have demonstrated its efficacy in high-risk patients with primary or secondary MR. Conventional TEER procedure, however, is performed under combined guidance of both echocardiography and fluoroscopy, which potentially results in high radiation exposure and limits its application. Since 2021 2021, the investigators have changed the procedural methodology by performing TEER under full echocardiographic guidance on accumulated dozens of MR patients successfully. To confirm the efficacy of a fully echo-guided TEER procedure, the investigators conduct the ECHO-CLIP study to compare its outcomes with the conventional TEER procedure, as well as evaluate the outcomes of this novel methodology in special populations with radiation contraindications. ECHO-CLIP study is a prospective, multicenter, open-label, noninferior, randomized controlled trial of TEER by two different methodological strategies in treating severe primary or secondary MR. It is anticipated to enroll a total of 200 patients as well to complete the enrollment before Dec 31, 2025 and the follow-up before Dec 31, 2026. This work will potentially demonstrate the feasibility and efficacy of the fully echo-guided TEER procedure, thereby revolutionizing the TEER methodology and benefiting more patients.

ELIGIBILITY:
Inclusion Criteria:

*Subjects meet either the first or second inclusion criteria in combination with the third and fourth ones were eligible.

1. Symptomatic DMR subjects with MR ≥ 3+ at high surgical risk in terms of STS Predicted Risk of Mortality replacement score ≥ 8 or STS Predicted Risk of Mortality repair score ≥ 6.*
2. FMR subjects with LVESD ≤ 70 mm and MR ≥ 3+, despite administration of GDMT for 30 days.*
3. MV anatomy appropriate for TEER procedure.
4. Subjects willing to participate in this study and complete the follow-up on schedule after obtaining informed consent.

Exclusion Criteria:

1. Myocardial infarction within 12 weeks prior to randomization.
2. Need for concurrent other cardiac procedures.
3. Any endovascular intervention or surgery within 30 days prior to randomization.
4. LVEF < 20%.
5. MV orifice area < 4.0 cm2.
6. Pulmonary artery systolic pressure > 70 mmHg, as determined by echocardiogram.
7. Severe mitral annular calcification.
8. Unsuitable MV anatomy potentially precluding clip implantation: leaflet calcification or significant leaflet cleft in the grasping zone.
9. Previous MV surgery or current implanted ventricular assist device or current implanted mechanical prosthetic valve.
10. Any intracardiac mass, thrombus, or vegetation, as evidenced by echocardiogram.
11. Active endocarditis or rheumatic heart disease.
12. History of DVT or PE.

Abbreviations: DMR, degenerative mitral regurgitation; MR, mitral regurgitation; STS, Society of Thoracic Surgeons; FMR, functional mitral regurgitation; LVESD, left ventricular end-systolic diameter; GDMT, guideline-directed medical therapy; TEER, transcatheter edge-to-edge repair; LVEF, left ventricular ejection fraction; MV, mitral valve; DVT, deep venous thrombosis; PE, pulmonary embolism.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-29 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
30-day successful rate after device implantation (residual MR ≤2+) | At 30 days after device implantation
  The primary outcome is the success rate of device implantation at 30 days ( residual MR≤moderate). Evaluation of the primary endpoints was done by specialized sonographers blinded to the intervention.

SECONDARY OUTCOMES:
1-year all-cause mortality | At 1 year after implantation
  All-cause mortality at 1 year after implantation.
1-year composite of death, reintervention, and recurrent MR ≥ 3+ | At 1 year after implantation
  Composite of death, reintervention, and recurrent MR ≥ 3+ at 1 year
Change in SF-36 score from baseline to 30 days and 1 year. | At 30 days and 1 year after implantation
  Change in 36-Item Short Form Survey score from baseline to 30 days and 1 year will be assessed. An increased score after implantation indicates an improvement in quality of life, while a decreased score after implantation indicates an impairment in quality of life.
Change in KCCQ score from baseline to 30 days and 1 year. | At 30 days and 1 year after implantation
  Change in Kansas City Cardiomyopathy Questionnaire score from baseline to 30 days and 1 year wiil be assessed. An increased score after implantation indicates an improvement in quality of life, while a decreased score after implantation indicates an impairment in quality of life.
Change in HADS score from baseline to 30 days and 1 year. | At 30 days and 1 year after implantation
  Change in Hospital Anxiety and Depression Scale score from baseline to 30 days and 1 year will be assessed. An increased score after implantation indicates an aggregation in psychological stress, while a decreased score after implantation indicates an improvement in psychological stress.
Composite of major adverse events | Immediately after implantation, at 30 days, 3 months, and at 1 year
  Composite of major adverse events immediately after implantation, at 30 days, 3 months, and at 1 year including death, myocardial infarction, reintervention, nonelective cardiovascular surgery for adverse events, ventilation over 48 hours, gastrointestinal complications requiring surgery, new-onset permanent atrial fibrillation, sepsis, and transfusion of 2 or more units of blood.
Left ventricular ejection fraction | At 30 days, 3 months, and 1 year after implantation
  Left ventricular ejection fraction at 30 days, 3 months, and 1 year
Left ventricular end-diastolic volume and left ventricular end-systolic volume | At 30 days, 3 months, and 1 year after implantation.
  Left ventricular end-diastolic volume and left ventricular end-systolic volume at 30 days, 3 months, and 1 year after implantation.
Left ventricular end-systolic diameter and left ventricular end-diastolic diameter | At 30 days, 3 months, and 1 year after implantation
  Left ventricular end-systolic diameter and left ventricular end-diastolic diameter at 30 days, 3 months, and 1 year after implantation
NYHA functional classification | At 30 days, 3 months, and 1 year after implantation.
  At 30 days, 3 months, and 1 year after implantation.
Regurgitant volume and regurgitant fraction | At 30 days, 3 months, and 1 year after implantation
  Regurgitant volume and regurgitant fraction at 30 days, 3 months, and 1 year.
Device implantation rate | At 30 days after device implantation
  Device implantation rate.
Vascular complications | At 30 days, 3 months, and 1 year after implantation
  Vascular complications at 30 days, 3 months, and 1 year including access-site hematoma > 6 cm, arteriovenous fistula, symptomatic peripheral ischemia or nerve injury with symptoms or signs over 48 hours, access-site vascular injury requiring surgical repair, PE, ipsilateral DVT, access-site associated infection requiring antibiotics injection or prolonging hospital stay.
Major bleeding events | At 30 days, 3 months, and at 1 year after implantation
  Major bleeding events at 30 days, 3 months, and at 1 year after implantation that is defined as any procedure-related bleeding requiring transfusion of 2 or more units of blood and/or surgical repair
Arrhythmia | At 30 days and 1 year after implantation
  Arrhythmia at 30 days, and at 1 year after implantation
Infective Endocarditis | At 30 days, 3 months and 1 year after implantation
  Infective Endocarditis at 30 days, 3 months, and at 1 year after implantation according to the Duke Criteria.
Thrombotic events | At 30 days, 3 months, and at 1 year after implantation
  Thrombotic events at 30 days, 3 months, and at 1 year after implantation.
Hemolytic events | At 30 days, 3 months, and at 1 year after implantation
  Hemolytic events at 30 days, 3 months, and at 1 year after implantation.
Iatrogenic atrial septal defect | At 30 days, 3 months, and at 1 year after implantation.
  Iatrogenic ASD at 30 days, 3 months, and at 1 year after implantation.
Single leaflet device attachment | At 30 days, 3 months, and at 1 year after implantation.
  Single leaflet device attachment at 30 days, 3 months, and at 1 year after implantation.
Mitral Stenosis | At 30 days, 3 months, and at 1 year after implantation.
  Mitral stenosis at 30 days, 3 months, and at 1 year after implantation that is defined as mitral valve area < 1.5 cm2.
Mitral valve area | At 30 days, 3 months, and at 1 year after implantation.
  Mitral valve area at 30 days, 3 months, and at 1 year after implantation.
Transmitral pressure gradient | At 30 days, 3 months, and at 1 year after implantation
  Transmitral pressure gradient at 30 days, 3 months, and at 1 year after implantation
Hospital stay after implantation | At study completion with an average of 1 year
  Hospital stay after implantation
ICU stay after implantation | At study completion with an average of 1 year
  ICU stay after implantation
30-day rehospitalization for heart failure | At 30 days after implantation
  Rehospitalization for heart failure at 30 days after implantation
New Warfarin Use | At 30 days and 1 year after implantation
  New Warfarin Use at 30 days and 1 year after device Implantation
Hospital cost | At study completion with an average of 1 year
  Hospital cost
Procedure time and radiation time | At study completion with an average of 1 year
  Procedure time and radiation time

CONTACTS AND LOCATIONS:
Overall Officials: Xiangbin Pan, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (1):
- Fuwai Hospital Chinese Academy of Medical Sciences Shenzhen, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ma J, Wang C, Wang S, Fang F, Zhang F, Yan X, Tang Y, Ouyang W, Pan X, Wang C. Design and Rationale of ECHO-CLIP Study: Transcatheter Edge-to-Edge Repair for Mitral Regurgitation Under Solely Transesophageal Echocardiographic Guidance Compared With Fluoroscopic and Transesophageal Echocardiographic Coguidance. J Am Heart Assoc. 2025 Jul;14(13):e040672. doi: 10.1161/JAHA.124.040672. Epub 2025 Jun 27. PMID 40576040